CLINICAL TRIAL: NCT02137434
Title: Influence of Dietary and Supplementary Calcium Over the Postprandial Effects of a Fatty Meal on Metabolism Profile, Blood Pressure, Oxidative Stress, and Endothelial Function of Obese Women.
Brief Title: Calcium Over Postprandial Effects of Fatty Meal on Metabolism, Blood Pressure, Oxidative Stress, Endothelial Function.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Antonio Felipe Sanjuliani, Associate Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: Acute calcium
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: Acute calcium; Dietary calcium; Supplementary calcium; Postprandial metabolism
MeSH Terms: conditions — Obesity | interventions — Calcium, Dietary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low calcium fatty meal (Placebo Comparator): Fatty meal consisting of biscuit, butter and drink made of albumin and sugar containing 40 mg of calcium, 600 kcal, with approximately 10% of energy from protein, 53% from fat, and 37% from carbohydrates.
- High dietary calcium fatty meal (Experimental): Fatty meal consisting of biscuit, butter and drink made of skimmed milk containing 540 mg of dietary calcium, 600 kcal, with approximately 10% of energy from protein, 53% from fat, and 37% from carbohydrates.
  Interventions: Other: Dietary calcium
- High supplementary calcium fatty meal (Experimental): Fatty meal consisting of biscuit, butter and drink made of albumin and sugar containing 540 mg of supplementary calcium from calcium carbonate, 600 kcal, with approximately 10% of energy from protein, 53% from fat, and 37% from carbohydrates.
  Interventions: Dietary Supplement: Supplementary calcium

INTERVENTIONS:
Other: Dietary calcium — Dietary calcium from skimmed milk
  Arms: High dietary calcium fatty meal
Dietary Supplement: Supplementary calcium — Supplementary calcium from calcium carbonate
  Arms: High supplementary calcium fatty meal

SUMMARY:
The purpose of the study is to investigate calcium acute influence over the postprandial effects of a fatty meal on serum calcium, plasma glucose and triglycerides, blood pressure, oxidative stress, and endothelial function in obese women.

DETAILED DESCRIPTION:
Studies suggest that dietary calcium intake is inversely associated with cardiovascular disease, but supplementary calcium appears to be associated with raised risk of cardiovascular events. Fatty meals lead to oxidative and inflammation which seems to interfere in postprandial dismetabolism, a predictor of cardiovascular events. To investigate calcium acute influence over the postprandial effects of a fatty meal a crossover, controlled, and randomized clinical trial will be conducted with obese adult women who will be randomized into one of the three interventions, characterized by a fatty meal with different contents of calcium: low calcium (40 mg), high dietary calcium (540 mg from non-fat milk), and high supplementary calcium (540 mg from calcium carbonate). Each participant will receive all three meals and one of them every week. Before meals' intake blood sample will be collected and endothelial function assess will be performed. Participants will eat the specific meal and endothelial function will be assessed again after 120 minutes. Blood sample collections will be repeated every 60 minutes after meal's intake to perform latter biochemical analyzes to determine: 8-isoprostane levels, to assess oxidative stress status; triglycerides; glucose; insulin; and serum calcium. Blood pressure will be continuously assessed during 25 minutes before meals' intake and during 2 hours after it.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) greater than or equal to 30 kg/m2 and below 40 kg/m2
* habitual dietary calcium intake below 500 mg per day

Exclusion Criteria:

* smoking
* dietary supplements or drugs that could interfere with body weight, metabolic profile and blood pressure
* diabetes
* thyroid dysfunction
* hypertension
* angina pectoris
* heart kidney or liver failure
* intestinal malabsorption
* acute or chronic inflammation
* HIV infection
* autoimmune diseases
* cancer
* chronic obstructive pulmonary disease
* dyslipidemia with indication for drug treatment
* history of myocardial infarction or stroke
* pregnancy and lactation
* menopause

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Blood pressure will be assessed continuously 25 min before meals' intake and 2 hours after it.
  Blood pressure will be assessed by digital photoplethysmography.

SECONDARY OUTCOMES:
Endothelial function | Endothelial function will be assessed after meals' intake and 2 hours after it.
  Endothelial function will be assessed by laser doppler fluxometry.

OTHER OUTCOMES:
Plasma triglycerides | Plasma triglycerides will be assessed in the fasting period and each hour during three hours after meals' intake
  Plasma triglycerides will be assessed by automated techniques
Plasma glucose | Plasma glucose will be assessed in the fasting period and each hour during three hours after meals' intake
  Plasma glucose will be assessed by glucose oxidase method.
Oxidative stress | Oxidative stress will be assessed in the fasting period and each hour during three hours after meals' intake
  Oxidative stress will be assessed by evaluating serum levels of 8-isoprostane and malondialdehyde by ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio F Sanjuliani, PhD., Principal Investigator — Discipline of Clinical and Experimental Pathophysiology, Rio de Janeiro State University
Locations (1):
- Discipline of Clinical and Experimental Pathophysiology, Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil